CLINICAL TRIAL: NCT02646085
Title: Multiparametric Imaging in Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yingbing Wang (Other)
Responsible Party: Sponsor-Investigator, Yingbing Wang, Radiologist, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015P001579
Record Dates: First submitted 2015-12-28; First posted 2016-01-05 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Methionine; 3-alpha-Hydroxysteroid Dehydrogenase (B-Specific)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): C11 Methionine positron emission tomography (PET/CT) studies will be performed as hybrid PET/CT examinations for attenuation correction and lesion localization. A bolus of 10 millicuries of C11 Methionine will be injected intravenously. Approximately 60 minutes following tracer injection, the patient will be positioned on a Siemens Biograph PET/CT scanner. A low milliampere CT of from the mid skull to mid thigh will be acquired first with while the patient is free breathing. PET will be acquired at 3 minutes per bed position using the 3D mode, approximately 6-7 bed positions. C11 Methionine PET/CT imaging will take less than 60 minutes.
  Interventions: Drug: C11 Methionine positron emission tomography

INTERVENTIONS:
Drug: C11 Methionine positron emission tomography — diagnostic positron emission tomography imaging after intravenous injection of C11 Methionine
  Other Names: L-methionine [C-11] methyl positron emission tomography

SUMMARY:
Patients with Multiple Myeloma will undergo single timepoint Positron Emission Tomography imaging with intravenously injected C11 Methionine to detect viable lesions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Myeloma with symptomatic bone or soft tissue disease
* Eastern Cooperative Oncology Group status 0 to 2
* Life expectance >= 12 weeks
* Ability to understand and willingness to sign informed consent
* Tissue sampling with genotype data planned within 3 months of C11 positron emission tomography (PET) imaging

Exclusion Criteria:

* Pregnant or breast feeding
* Claustrophobic reactions and unable to lie still on a bed inside the PET scanner for 60 minutes
* Research related radiation exposure exceeding 50 millisieverts

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Quantitative measure of C11 Methionine uptake | 12 months
  Standardized uptake value (a semiquantitative, unit less measure of radioactivity normalized for injected activity and body weight) will be measured for individual C11 Methionine uptake abnormalities (defined as focally increased uptake higher than background levels in a similar tissue type). All abnormal uptake not in locations common for benign etiologies, such as fracture and degenerative change, will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Wang Y, Yee A, Bernstein Z, O'Donnell E, Raje N, Mahmood U. Carbon-11-Labeled Methionine PET/CT in Patients With FDG-Occult Multiple Myeloma: A Prospective Pilot Study. AJR Am J Roentgenol. 2023 Apr;220(4):578-579. doi: 10.2214/AJR.22.28560. Epub 2022 Nov 16. PMID 36382911